CLINICAL TRIAL: NCT03972475
Title: A Multi Center Observational Study on the Effects of Maintenance Fluids on Overall Fluid Balance in ICU Patients.
Brief Title: The Effect of Maintenance Fluids on Overall Fluid Balance in ICU Patients
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/
Record Dates: First submitted 2019-05-24; First posted 2019-06-03 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Fluid Overload; Fluid Therapy; Critical Care
MeSH Terms: conditions — Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Biospecimen Retention: None Retained — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The amount of fluids characterized as non-resuscitation fluids given to ICU patients are likely to be high and will probably have a substantial impact on the total amount of fluid administered to ICU patients daily. It will most likely also influence on the total fluid balance and the negative outcome of fluid overload.

The aim of our study is to investigate the amount of fluid given as maintenance fluids in the ICU and the impact of this fluid on total fluid balance.

DETAILED DESCRIPTION:
Fluid therapy is an important part in both prevention and treatment of shock and multiple organ dysfunction in the ICU. However, the risks of giving patients too much fluids resulting in fluid has been gaining increased focus during recent years. Numerous studies regarding the amount of resuscitation fluid given to ICU patients have been performed, as well as investigations regarding factors that trigger the decision to deliver a fluid challenge to the patients. Likewise, multiple studies reveal that a more restrictive use of resuscitation fluids often lead to a better outcome for our patients.

However, data regarding the amount of maintenance fluids and the effect of maintenance fluids on fluid balance and consequently outcome remain sparse. One major difficulty is that there is no universal definition of the term maintenance fluid. Some researchers include all fluids that is not considered resuscitation fluids, i.e. fluids given to administer drugs, to keep peripheral and central venous catheters functioning, administration of basal fluid needs and nutrition, while others exclude fluids covering basal needs and nutrition from the definition.

ELIGIBILITY:
Inclusion Criteria: All ICU patients that spent one week or more in the ICU. -

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that spend one week or more in the general ICUs at the included hospitals. Data will be collected from day 3 of the ICU stay until day 7.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
Fluid balance | One week
  To register the volume of fluid given to ICU patients categorized as resuscitation fluid, fluid to cover basal needs and nutrition and as fluid given to administer drugs and keeping intravenous accesses functioning. This will be measured i milliliters of fluid that the patients receive intravenously and orally by studying patient charts manually from their stay in the ICU.

SECONDARY OUTCOMES:
Fluid needs vs actual fluids given | One week
  To relate the quantity of maintenance fluid given to the patients with their theoretical fluid needs, by counting their needs (basal need of 30 mls/kg/day, previous losses and ongoing losses) and comparing it to the amount of fluid that the patient has actually received (by going through patient charts from their ICU stay).
Electrolyte | One week
  Total amount of electrolytes given to the patients intravenously or orally in the study, measured in mmol, by manually going through charts from patients ICU-stay.

CONTACTS AND LOCATIONS:
Overall Officials: Miklos Lipcsey, Assoc prof, Study Director — Uppsala University
Locations (6):
- Sweden (6):
  - ICU, Karolinska Hospital Huddinge, Huddinge, Stockholm County
  - ICU, Karolinska hospital Solna, Solna, Stockholm County
  - ICU, Mälarsjukhuset Eskilstuna, Eskilstuna
  - ICU, Gävle Hospital, Gävle
  - ICU, Sahlgrenska University Hospital, Gothenburg
  - Central ICU (CIVA), Uppsal university hospital, Uppsala

REFERENCES:
- [Derived] Nihlen S, Frithiof R, Titze J, Kawati R, Rasmusson J, Rylander C, Pikwer A, Castegren M, Belin A, Hultstrom M, Lipcsey M. The Contribution of Plasma Urea to Total Osmolality During Iatrogenic Fluid Reduction in Critically Ill Patients. Function (Oxf). 2021 Oct 29;3(1):zqab055. doi: 10.1093/function/zqab055. eCollection 2022. PMID 35330925
- [Derived] Nihlen S, Kawati R, Rasmusson J, Rylander C, Pikwer A, Castegren M, Belin A, Lipcsey M. Hidden sources of fluids, sodium and potassium in stabilised Swedish ICU patients: A multicentre retrospective observational study. Eur J Anaesthesiol. 2021 Jun 1;38(6):625-633. doi: 10.1097/EJA.0000000000001354. PMID 33074941